CLINICAL TRIAL: NCT06701266
Title: Diagnostic Agreement of Human Interleukin-6 Chairside Point-of-Care Test (PoCT) to Enzyme-Linked Immunosorbent Assay (ELISA) in Teeth with Apical Periodontitis
Brief Title: Accuracy of PoCT to ELISA by Detecting Human IL-6 in Teeth with Apical Periodontitis
Acronym: PoCT ELISA
Status: Not yet recruiting | Type: Observational
Sponsor: Manipal University College Malaysia (Other)
Collaborators: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Dr. Anchu Rachel Thomas, Associated Professor of Conservative Dentistry & Endodontics, Melaka Manipal Medical College
Other Study IDs: MUCM/005D/11/2024
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient have apical periodontitis: Patient have single rooted tooth with apical periodontitis that undergo RCT in MUCM.
  Interventions: Device: Point of Care Test

INTERVENTIONS:
Device: Point of Care Test — PoCT as a chairside test, ELISA as a gold standard

SUMMARY:
To compare the diagnostic agreement of human IL-6 chairside PoCT to ELISA in apical periodontitis undergoing endodontic therapy which could be clinically helpful to monitor the healing of periapical tissues enabling the clinician to complete the endodontic procedure, leading to a better patient care.

This study will be conducted at the Conservative and Endodontics Department in Polyclinic B, Faculty of Dentistry, Manipal University College Malaysia (MUCM). It involves 30 selected patients who have single rooted tooth with apical periodontitis that undergo RCT. The collection of the exudate from the canal will be on pre and post-instrumentation. The exudated will collect twice in each instrumentation for PoCT and ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Patient having single root tooth with AP that is negative to the pulp sensitivity test
* Presence of periapical lesion

Exclusion Criteria:

* Pregnancy

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who is having apical periodontitis and undergo RCT in MUCM
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Detect the IL-6 in the exudate of the tooth with apical periodontitis | 1 week
  Collection of exudate in Pre-instrumentation for PoCT and ELISA . After 1 week, collection of exudate in post-instrumentation for PoCT and ELISA will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Manipal University College Malaysia, Malacca, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: No